CLINICAL TRIAL: NCT05670873
Title: Effect of Individual Biofeedback Transcranial Magnetic Stimulation Assessed by a Hybrid Neural Network Evaluation Model on Disorder of Consciousness in Acute Severe Cerebrovascular Disease Patients
Brief Title: Transcranial Magnetic Stimulation in Disorder of Consciousness in Acute Severe Cerebrovascular Disease Patients
Acronym: I-HELP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liping Liu (Other)
Responsible Party: Sponsor-Investigator, Liping Liu, Professor, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-HELP
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Stroke; Consciousness Disorder; Transcranial Magnetic Stimulation
Keywords: Ischemic Stroke; Consciousness Disorder; Transcranial Magnetic Stimulation; Hybrid Neural Network Evaluation Model
MeSH Terms: conditions — Ischemic Stroke; Consciousness Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS treatment (Experimental): 20 days of repetitive transcranial magnetic stimulation: stimulation site is the left dorsolateral prefrontal cortex, stimulation intensity at 90% RMT, stimulation frequency is 10Hz. A total of 1000 pulses, 10s 10Hz train stimulation, repeated 10 times, each interval 60s, a total of 11 minutes and 40 seconds, 1 treatment per day, a total of 20 days.
  Interventions: Device: Transcranial magnetic stimulation
- iTBS treatment (Experimental): 20 days of intermittent theta-burst stimulation: stimulation site is the left dorsolateral prefrontal cortex, stimulation intensity at 90% RMT, stimulation frequency is 50Hz. A total of 600 pulses, 3 pulses each time, with an interval of 200 ms, for a total of 2 seconds (10 groups), and then repeat the above process after an interval of 10 seconds, a total of 190 seconds, 1 treatment per day, a total of 20 days.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial magnetic stimulation given to the left dorsolateral prefrontal cortex

SUMMARY:
This study is aimed at evaluating the potential of transcranial magnetic stimulation in patients with acute severe ischemic stroke with DoC while assessing patients with a hybrid neural network evaluation model. This model may be the basis for initiating individualized closed-loop neuromodulation treatment in patients with DoC.

DETAILED DESCRIPTION:
Despite continued advances in life-sustaining intensive care for severe brain injury patients, little can be done to promote behavioral recovery in patients with disorder of consciousness (DoC). Arousal is the primary task in the rehabilitation of patients with impaired consciousness. Evidence suggests that some medications and physical therapies can induce wakefulness by reactivating specific pathways that lead to impaired consciousness. However, due to the complexity of the type, degree, location, and other related influencing factors of brain injury, the current commonly used treatment options are not effective for patients with impaired consciousness, and the theoretical basis for benefit is not sufficient.

This study is aimed at evaluating the potential of transcranial magnetic stimulation in patients with acute severe ischemic stroke with DoC while assessing patients with a hybrid neural network evaluation model. This model may be the basis for initiating individualized closed-loop neuromodulation treatment in patients with DoC.

Before and after a course of treatment (20 days), activation and connectivity of patients' arousal centers will be assessed through a hybrid neural network evaluation model, which consists of comprehensive cortical connectivity parameters (perturbational complexity index and evoked high-frequency oscillations) and region-specific cortical connectivity parameters (short-latency afferent inhibition and mismatch negativity). Each parameter is clinically used to assess a patient's level of cortex connectivity. This hybrid evaluation model may give a comprehensive evaluation of a patient's degree of awareness, and enhance our understanding of the mechanisms underlying these conditions.

ELIGIBILITY:
Inclusion Criteria:

* 7-28 days after ischemic stroke
* behavioral profile consistent with a UWS or MCS as assessed with the Coma Recovery Scale Revise
* prestroke Modified Ranking Scale(mRS) ≤2

Exclusion Criteria:

* history of vascular malformation or aneurysmal SAH or untreated aneurysm prior to stroke
* disorder of consciousness prior to stroke
* impairment of hearing
* metal implants, e.g. stenting, pacemaker, etc.
* contraindications to MRI, such as claustrophobia
* history of epilepsy or epileptic episodes
* suffering from serious diseases such as malignant tumors, etc., with expected survival time <1 year
* patient is currently involved with other trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale Revised (CRS-R) | Change in maximum CRS-R score from baseline to 1 month
  The Coma Recovery Scale Revised (CRS-R) is a standard clinical protocol specifically developed to assess a patient's level of consciousness, and does so by evaluating a patient's level of responsiveness to sensory stimulation, their ability to understand language, and to communicate. This procedure is typically administered at bedside. The protocol is divided into 6 sub-scales, each assessing a different area (e.g., visual function, auditory function, communication, arousal), and the final score is calculating by adding all sub-scales.The total score of this scale goes from its minimum, 0, which implied a state of coma, to 23, which implies emergence from a Minimally Conscious State (i.e., eMCS). Higher values thus map onto better outcomes.
Number of Participants With (Severe) Adverse Events | day 20 (+/-3)
  Number of AEs and SAEs occurring throughout the paradigm.

SECONDARY OUTCOMES:
Hybrid Neural Network Evaluation | Change from baseline to day 20 (+/-3)
  The Hybrid Neural Network Evaluation Model consists of comprehensive cortical connectivity parameters (perturbational complexity index and evoked high-frequency oscillations) and region-specific cortical connectivity parameters (short-latency afferent inhibition and mismatch negativity). Each parameter is clinically used to assess a patient's level of cortex connectivity. This hybrid evaluation model may give a comprehensive evaluation of a patient's degree of awareness, and enhance our understanding of the mechanisms underlying these conditions
Number of voxels in which the Functional Magnetic Resonance Imaging (fMRI) signal is significantly associated to TMS across the whole group | Change from baseline to 1 month
  Number of voxels found to have a functional MRI signal (measured with a Blood Oxygenation Level Dependent sequence) significantly associated with the TMS stimulation across the tested population.

CONTACTS AND LOCATIONS:
Overall Officials: Liping Liu, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No